CLINICAL TRIAL: NCT03416803
Title: Prediction of Lymph Node Metastasis in Hepatocellular Carcinoma and the Study of Individualized Radiotherapy
Brief Title: A Study of Individualized Radiotherapy Based on a Prediction Model of Lymph Node Metastasis in Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZS-LNM-2017
Record Dates: First submitted 2018-01-08; First posted 2018-01-31 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Lymph Node Metastasis; Hepatocellular Carcinoma; Radiotherapy
MeSH Terms: conditions — Lymphatic Metastasis; Carcinoma, Hepatocellular | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy (Experimental): Patients in the experimental group, who were at high risk for lymph node metastasis, underwent radiotherapy in the lymphatic drainage area. Radiotherapy was started in lymphatic drainage areas about 1 month after HCC surgery. The range of radiotherapy was hepatic portal area, pancreas circumference, celiac trunk and abdomen Around the aortic lymph drainage area, the dose of radiation 45Gy, conventional segmentation.
  Interventions: Radiation: Radiotherapy
- Blank control (No Intervention): Patients in the control group , who were at high risk for lymph node metastasis，were followed up.

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy
  Arms: Radiotherapy

SUMMARY:
Objectives:

1. To further validate the predictive efficacy of our established microRNA prediction model of HCC lymph node metastasis.
2. To establish a precise therapeutic mode of prophylactic radiation therapy in high-risk patients with HCC with lymph node metastasis under the guidance of a microRNA prediction model.

DETAILED DESCRIPTION:
First, screening out patients who underwent hepatic tumor resection and pathologically diagnosed as HCC .

Then，performing the detection of miR-145, miR-31 and miR-92a by using the HCC lymph node metastasis microRNA correlation prediction model established in our previous study. The patients are judged as high risk of lymph node metastasis and low risk Patients, then high-risk patients under the condition of informed consent into the group, randomized into treatment group and control groups.

Last, Patients enrolled in the treatment group were treated with radiotherapy and followed up.

ELIGIBILITY:
Inclusion Criteria:

1. patients underwent liver tumor resection and pathological diagnosis of HCC in our hospital.
2. The tumor samples of these HCC patients were detected by in situ hybridization with miR-145, miR-31 and miR-92a. We used the previously established HCC lymph node metastasis microRNA prediction model to determine the patients with high-risk lymph node metastasis and low-risk patients at high risk Patients were randomly assigned into treatment group and control group with informed consent.
3. HCC patients were not receive other anti-cancer treatment.
4. Blood routine examination was normal.
5. Child-Pugh grade A, normal liver and kidney function in the normal range (including ALT or ASL within 2.5 times the normal), WBC> 3 × 109 / L, Hb> 90g / L, PLT> 50 × 109 /
6. HCC patients were not receive the history of upper abdominal radiotherapy.
7. sign the informed consent.
8. age 18-75 years old.
9. KPS score 80-100 points.

Exclusion Criteria:

1. accepted other anti-cancer treatment.
2. Patients was determined to be low-risk lymph node metastasis by the pre-established HCC lymph node metastasis microRNA prediction model.
3. blood and liver and kidney dysfunction.
4. can not control the infection.
5. at the same time the merger of other malignant tumors.
6. while using other experimental drugs or to participate in other clinical trials.
7. serious heart, lung, kidney disease.
8. pregnant or lactating women.
9. serious nervous system disease, can not clearly tell the treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival | The outcome measures are assessed up to 2 years.
  The therapeutic effects are mainly evaluated by the 2-year overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongshan Hospital, PhD, Principal Investigator — Fudan University, Shanghai,China
Locations (1):
- 180 Fenglin Road, Shanghai, China